CLINICAL TRIAL: NCT06061094
Title: A Multicentre, Randomized Trial in Adults With de Novo Philadelphia-Chromosome Positive Acute Lymphoblastic Leukemia to Assess the Efficacy of Ponatinib Versus Imatinib in Combination With Low-intensity Chemotherapy, to Compare End of Therapy With Indication for SCT Versus TKI, Blinatumomab and Chemotherapy in Optimal Responders and to Evaluate Blinatumomab in Suboptimal Responders (GMALL-EVOLVE)
Brief Title: Randomized Trial in Adult de Novo Ph Positive ALL With Chemotherapy, Imatinib or Ponatinib, Blinatumomab and SCT
Acronym: GMALL-EVOLVE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Deutsche Leukämie- & Lymphom-Hilfe (Unknown); German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Nicola Goekbuget, Dr. Nicola Gökbuget, Goethe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMALL-EVOLVE; 2022-000760-21 (EudraCT Number)
Record Dates: First submitted 2023-08-20; First posted 2023-09-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-09

CONDITIONS: Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia
Keywords: Philadelphia Chromosome Positive Acute Lymphoblastic Leukemia; Tyrosinekinase Inhibitors; Blinatumomab
MeSH Terms: interventions — Imatinib Mesylate; ponatinib; blinatumomab; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- A: Imatinib + low dose chemotherapy (Active Comparator): Imatinib 600mg QD + low dose chemotherapy induction and consolidation I (Standard Arm of Randomization I)
  Interventions: Drug: Imatinib
- B: Ponatinib + low dose chemotherapy (Experimental): Ponatinib 45mg QD (reduction to 30mg QD after Induction) + low dose chemotherapy induction and consolidation I (Experimental Arm of Randomization I)
  Interventions: Drug: Ponatinib
- C: Molecular CR: End of therapy with indication for SCT (Active Comparator): Molecular CR: End of therapy with indication for SCT (Standard Arm of Randomization II)
  Interventions: Other: Indication for stem cell transplantation
- D: Molecular CR: continuation with Imatinib/Ponatinib (per Rando I), chemotherapy and Blinatumomab (Experimental): Molecular CR: No end of therapy with indication for SCT but and continuation with Imatinib/Ponatinib (per Randomization I), chemotherapy and Blinatumomab (Experimental Arm of Randomization II)
  Interventions: Drug: Imatinib; Drug: Ponatinib; Drug: Blinatumomab
- E: Mol Fail / Mol NE: Continuation with Imatinib/Ponatinib (per Rando I) and addition of Blina (Experimental): Molecular Failure / Molecular Not Evaluable: Continuation with Imatinib/Ponatinib (per Randomization I) and addition of Blinatumomab (Experimental Arm)
  Interventions: Drug: Imatinib; Drug: Ponatinib; Drug: Blinatumomab; Other: Indication for stem cell transplantation

INTERVENTIONS:
Drug: Imatinib — Imatinib 600mg QD plus Chemotherapy
  Arms: A: Imatinib + low dose chemotherapy; D: Molecular CR: continuation with Imatinib/Ponatinib (per Rando I), chemotherapy and Blinatumomab; E: Mol Fail / Mol NE: Continuation with Imatinib/Ponatinib (per Rando I) and addition of Blina
Drug: Ponatinib — Ponatinib 45 mg QD plus chemotherapy
  Arms: B: Ponatinib + low dose chemotherapy; D: Molecular CR: continuation with Imatinib/Ponatinib (per Rando I), chemotherapy and Blinatumomab; E: Mol Fail / Mol NE: Continuation with Imatinib/Ponatinib (per Rando I) and addition of Blina
Drug: Blinatumomab — Patients with molecular failure or intermediate response receive one cycle Blinatumomab before SCT; Patients with molecular CR randomized to the experimental arm receive 3 cycles Blinatumomab + chemotherapy
  Arms: D: Molecular CR: continuation with Imatinib/Ponatinib (per Rando I), chemotherapy and Blinatumomab; E: Mol Fail / Mol NE: Continuation with Imatinib/Ponatinib (per Rando I) and addition of Blina
Other: Indication for stem cell transplantation — Patients with molecular CR randomized to the standard arm have an indication for SCT; patients with molecular failure or intermediate response have an indication for SCT. SCT is not part of the trial.
  Arms: C: Molecular CR: End of therapy with indication for SCT; E: Mol Fail / Mol NE: Continuation with Imatinib/Ponatinib (per Rando I) and addition of Blina

SUMMARY:
The current Standard of Care (SoC) in younger patients with Ph+ ALL is Imatinib in combination with low-dose chemotherapy, change of TKI in case of persistent MRD above 10-3 after consolidation I and indication for stem cell transplantation.

The EVOLVE trial aims to answer three questions challenging the current SoC:

Use of Ponatinib compared to Imatinib both in combination with low-dose chemotherapy and consolidation I (randomization I).

In MRD good responders: Omit end of therapy in primary care and indication for SCT but continue therapy with TKI, chemotherapy and Blinatumomab as additional antileukemic compound (randomization II).

In MRD poor responders: Omit indication for TKI change but give instead Blinatumomab followed by end of therapy in primary care and indication for SCT (non-randomized).

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients >= 18 years, <=65 years
* Philadelphia chromosome or BCR-ABL1 positive ALL
* Not previously treated except with corticosteroids ≤ 7 days, standard GMALL prephase with dexamethasone and cyclophosphamide including intrathecal therapy, hydroxyurea, a single dose vincristine or other cytostatic drugs and start of standard induction for Ph-positive ALL (1 dose vincristine, 1 dose of Rituximab, 2 doses dexamethasone and up to 5 days Imatinib)
* ECOG performance status ≤2
* Signed written inform consent
* Molecular evaluation for BCR-ABL1 performed
* Negative pregnancy test in women of childbearing potential
* Woman of childbearing potential willing to use 2 highly effective methods of contraception while receiving study treatment and for an additional 3 months after the last dose of study treatment (Pearl-Index <1%). Male who has a female partner of childbearing potential willing to use 2 highly effective forms of contraception while receiving study treatment and for at least an additional 3 months after the last dose of study treatment (Pearl-Index <1%).
* Normal serum levels > LLN (lower limit of normal) of potassium and magnesium, or corrected to within normal limits with supplements, prior to the first dose of study medication
* Serum lipase ≤ 1.5 x ULN. For serum lipase > ULN - ≤ 1.5 x ULN, value must be considered not clinically significant and not associated with risk factors for acute pancreatitis
* Normal QTcF interval ≤450 ms for males and ≤470 ms for females
* Signed and dated written informed consent is available
* Participation in the registry of the German Multicenter Study Group for Adult ALL (GMALL)

Exclusion Criteria:

* History of malignancy other than ALL diagnosed within 5 years (yrs) prior to start of protocol-specified therapy with defined exceptions
* Contraindications against the use of Imatinib, Ponatinib, chemotherapy or Blinatumomab
* Patient previously treated with tyrosine kinase inhibitors
* Nursing women
* Known impaired cardiac function, including any of the following: as detailed in protocol
* Symptomatic peripheral vascular disease
* Any history of ischemic stroke or transient ischemic attacks (TIAs)
* Uncontrolled hypertriglyceridaemia
* History or presence of clinically relevant CNS pathology as detailed in protocol
* History or active relevant autoimmune disease
* Known hypersensitivity to immunoglobulins or to any other component of the study drug formulation
* Known diagnosis of human immunodeficiency virus (HIV) infection (HIV testing is not mandatory) or active infection with Hepatitis B or C
* History of pancreatitis within 6 months previous to start of treatment within the trial
* Treatment with any other investigational agent or participating in another trial within 30 days prior to entering this study
* Inadequate hepatic functions defined as ASAT or ALAT > 2,5 times the institutional upper limit of normal or > 5 times ULN if considered due to leukemia
* Total bilirubin > 1.5-fold the institutional upper limit unless considered to be due to organ involvement by the leukemia or to M. Gilbert / M. Meulengracht
* Concurrent severe diseases which exclude the administration of therapy e.g. severe, uncontrolled acute or chronic infections
* Inability to understand and/or unwillingness to sign a written informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-07-14 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
OS in MolCR patients treated with TKI-Chemo-Blina versus (vs) EOT with indication for SCT (Standard of Care) | up to 4 years from randomization I
  Probability of overall survival up to 4 years from randomization I in patients with mo-lecular remission after consolidation 1 comparing a combination treatment of TKI, Blina-tumomab and chemotherapy versus EOT with indication for SCT

SECONDARY OUTCOMES:
Rate of molecular complete remission at week 11 after consolidation | week 11 after consolidation
  Rate of molecular complete remission at week 11 after consolidation with chemotherapy in combination with Ponatinb versus Imatinib

OTHER OUTCOMES:
Probability of remission duration | at 2 years, 3 years, 4 yrs
  Probability of remission duration
Cumulative incidence of relapse | at 2 years, 3 years, 4 yrs
  Cumulative incidence of relapse
Mortality in CR | at 2 years, 3 years, 4 yrs
  Mortality in CR
Probability of relapse-free survival | at 2 years, 3 years, 4 yrs
  Probability relapse-free survival
Hematologic/Molecular response | after induction I (3 weeks), after induction II (6 weeks) and after consolidation I (11 weeks)
  Proportion of patients who achieve hematological and molecular remission or experience molecular failure
Overall incidence and severity of AEs | during induction therapy (approximately 6 weeks)
  Overall incidence and severity of AEs in patients (CTC-AE 4.0) receiving ponatinib versus imatinib during induction therapy
Probability of continuous molecular remission | at 2, 3 and 4 yrs
  Probability of continuous molecular remission at different time-points of Ponatinib versus Imatinib-based therapy
Measuring log-reduction (kinetic on MRD response) | after induction I (3 wks), after induction II (6 wks) and after consolidation I (11 wks)
  Measuring log-reduction (kinetic on MRD response) in patients with a Ponatinib versus Imatinib-based therapy
Probability of MRD response including the induction of complete molecular remission and measurement the log-reduction of MRD | after induction I (3 weeks), after induction II (6 weeks) and after consolidation I (11 weeks)
  Probability of MRD response including the induction of complete molecular remission and measurement the log-reduction of MRD in patients with blinatumomab in combination with Ponatinib versus Imatinib in patients with molecular persistence (molecular failure and MRD positivity below quantitative range) after consolidation 1
Probability of continuous MRD response and molecular remission and duration of molecular remission | After consolidation 1 approximately every three months
  Probability of continuous MRD response and molecular remission and duration of molecular remission at different time-points in patients with molecular persistence (molecular failure and not quantifiable) receiving Blinatumomab in combination with Ponatinib versus Imatinib after consolidation 1
Overall incidence and severity of AEs in patients | during each treatment cycle
  Overall incidence and severity of AEs in patients (CTC-AE 4.0) receiving Ponatinib or Imatinib in combination with Blinatumomab and chemotherapy
Probability of continuous MRD response | at 2, 3 and 4 years
  Probability of continuous MRD response and molecular remission and duration of molecular remission at different time-points in patients with Blinatumomab in combination with Ponatinib and chemotherapy or Imatinib and chemotherapy and rate of molecular relapse
Time to molecular remission | after induction I (3 weeks), after induction II (6 weeks) and after consolidation I (11 weeks)
  Time to molecular remission measured by time-point of first achievement
Incidence of TKI dose reductions | for each cycle - approximately 28 days each - number of cycles depends on treatment arm
Incidence of TKI changes | for each cycle - approximately 28 days each - number of cycles depends on treatment arm
Incidence of TKI treatment interruptions | for each cycle - approximately 28 days each - number of cycles depends on treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Goekbuget, MD, Principal Investigator — Department of Medicine, Hematology and Oncology, Goethe University Frankfurt, Frankfurt, Germany; Fabian Lang, MD, Principal Investigator — Department of Medicine, Hematology and Oncology, Goethe University Frankfurt, Frankfurt, Germany; Heike Pfeifer, MD, Principal Investigator — Department of Medicine, Hematology and Oncology, Goethe University Frankfurt, Frankfurt, Germany
Locations (85):
- Germany (85):
  - Uniklinik RWTH Aachen, Aachen
  - Klinikum Aschaffenburg, Aschaffenburg
  - Klinikum Augsburg, Augsburg
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Klinikum Bayreuth, Bayreuth
  - Vivantes Klinikum am Urban, Berlin
  - Charité Universitätsmedizin Berlin, Berlin
  - Vivantes Klinikum Neukölln, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Charite Berlin Virchow Klinikum, Berlin
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - UK Knappschaftskrankenhaus Bochum, Bochum
  - Evangelische Kliniken Bonn, Bonn
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte, Bremen
  - Klinikum Chemnitz, Chemnitz
  - Universitätsklinikum Köln, Cologne
  - Klinikum Darmstadt, Darmstadt
  - Städtisches Klinikum Dessau, Dessau
  - Klinikum Dortmund, Dortmund
  - St. Johannes Hospital Dortmund, Dortmund
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
  - Helios Klinikum Duisburg, Duisburg
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Marien Hospital Düsseldorf, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - St.-Antonius-Hospital, Eschweiler
  - Universitätsklinikum Essen, Essen
  - Evangelisches Krankenhaus Essen-Werden, Essen
  - Department of Medicine, Hematology and Oncology, Goethe University Hospital Frankfurt, Frankfurt
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Niels-Stensen-Kliniken Georgsmarienhütte, Georgsmarienhütte
  - Wilhelm-Anton-Hospital, Goch
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Klinikum Gütersloh, Gütersloh
  - Katholisches Krankenhaus Hagen, Hagen
  - Universitätsklinikum Halle, Halle
  - Asklepios Klinik St. Georg Hamburg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Marien Hospital Herne, Herne
  - Universitätsklinikum des Saarlandes, Homburg
  - Klinikum Idar-Oberstein, Idar-Oberstein
  - Universitätsklinikum Jena, Jena
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - St. Vincentius-Kliniken Karlsruhe, Karlsruhe
  - Klinikum Kassel, Kassel
  - Universitätsklinikum Kiel, Kiel
  - Gemeinschaftsklinikum Mittelrhein, Koblenz
  - Universitätsklinikum Leipzig, Leipzig
  - Märkische Kliniken Lüdenscheid, Lüdenscheid
  - Universitätsklinikum Magdeburg, Magdeburg
  - UNIVERSITÄTSMEDIZIN der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinikum Mannheim, Mannheim
  - Philipps-Universität Marburg, Marburg
  - Kliniken Maria Hilf Möchengladbach, Möchengladbach
  - LMU Klinikum München, München
  - Klinikum Rechts der Isar TU München, München
  - Universitätsklinikum Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - Ortenau Klinikum Offenburg, Offenburg
  - Klinikum Oldenburg, Oldenburg
  - Brüderkrankenhaus St. Josef Paderborn, Paderborn
  - Klinikum Passau, Passau
  - Klinikum Ernst von Bergmann, Potsdam
  - Krankenhaus Barmherzige Brüder Regensburg, Regensburg
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Rostock, Rostock
  - Agaplesion Diakonieklinikum Rotenburg, Rotenburg (Wümme)
  - Diakonie-Krankenhaus Schwäbisch-Hall, Schwäbisch Hall
  - Katharinenhospital Stuttgart, Stuttgart
  - Diakonissenkrankenhaus Stuttgart, Stuttgart
  - Robert-Bosch-Krankenhaus Stuttgart, Stuttgart
  - Klinikum Traunstein, Traunstein
  - Mutterhaus der Borromäerinnen Trier, Trier
  - Krankenhaus d. Barmherzigen Brüder, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm
  - Klinikum Schwarzwald-Baar, Villingen-Schwenningen
  - Helios Klinikum Wuppertal, Wuppertal
  - Universitätsklinikum Würzburg, Würzburg
  - Heinrich-Braun Klinikum, Zwickau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Lang et al, Oncol Res Treat 2024;47:430-433 — https://pubmed.ncbi.nlm.nih.gov/38754400/